CLINICAL TRIAL: NCT02779322
Title: Prospective Randomized Controlled Clinical Trial: Laparoscopic Roux-en-Y Gastric Bypass Versus Laparoscopic One Anastomosis Gastric Bypass
Brief Title: Laparoscopic Roux-en-Y Gastric Bypass Versus Laparoscopic One Anastomosis Gastric Bypass
Acronym: OAGB-vs-LRYGB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Puerta de Hierro University Hospital (Other)
Responsible Party: Principal Investigator, Miguel J. Garcia-Oria, MD, PhD, Puerta de Hierro University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06082015
Record Dates: First submitted 2016-05-16; First posted 2016-05-20 (Estimated); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Morbid Obesity; Postoperative Complications; Weight Loss
Keywords: gastric bypass; hospital charges; mini gastric bypass
MeSH Terms: conditions — Obesity, Morbid; Postoperative Complications; Weight Loss | interventions — Single Person; Gastric Bypass

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Minigastric bypass (Active Comparator): Intervention(s): The patient will have done a Laparoscopic one anastomosis gastric bypass (minigastric bypass) at the time of the surgical procedure.
  Interventions: Procedure: Minigastric bypass
- Gastric bypass (Active Comparator): The patient will have a Laparoscopic Roux-en-Y gastric bypass at the time of the surgical procedure
  Interventions: Procedure: Gastric bypass

INTERVENTIONS:
Procedure: Minigastric bypass — The patient will be submitted to a minigastric bypass at the time of the operation
  Other Names: Single or One anastomosis gastric bypass
  Arms: Minigastric bypass
Procedure: Gastric bypass — In this case a simplified conventional gastric bypass will be performed
  Other Names: Laparoscopic gastric bypass
  Arms: Gastric bypass

SUMMARY:
This study try to identify differences in cost, length of operation and results between two different bariatric surgical techniques, the laparoscopic Roux-en-Y gastric bypass and the Single anastomosis laparoscopic gastric bypass. The study will be conducted in a Spanish public health system hospital.

The patients of the trial will have the preoperative studies, hospital treatment during the admission, postoperative treatment and follow up as any other patient included in the hospital bariatric surgery program. No new methods are applied other than randomly choose the surgical technique.

Patients will be randomized in a 1:1 ratio to each group.

DETAILED DESCRIPTION:
One group of patients of the study will have done the simplified laparoscopic gastric bypass, with a vertical gastric pouch of about 20 ml, a 150 cm Roux-en-Y limb constructed in an antegastric antecolic fashion, and a biliary limb of 100 cm. Anastomosis will be done with endoscopic surgical linear stapler, closing the apertures with continuous absorbable running sutures. The Petersen space and the mesenteric defect will be closed with non-absorbable sutures.

The other group of patients will have performed the single anastomosis gastric bypass, also known as the Minigastric bypass (MGB), which have a vertical gastric pouch about 100-150 ml, and an end to side gastro-jejunal anastomosis at 200 cm from Treitz angle. The anastomosis will be done with endoscopic surgical linear stapler, closing the aperture with continuous absorbable running sutures.The Petersen space will be also close with non-absorbable sutures.

The investigators randomly assigned 10 patients to each group, n=20. Considering that one of the methods is basically the same than the other, but for the Roux-en-Y construction, it is expected a clear difference in operating room (OR) time, between groups. Fisher Test, will be used for the statistical analysis, assuming a risk of 0.05 and a statistical power of 90%, and Mann-Whitney test for quantitative parameters.

Once patients were included in the study, they were randomized in a 1:1 ratio to the conventional laparoscopic gastric bypass group or the single-anastomosis laparoscopic gastric bypass (Mini gastric bypass) group and were also blinded to the surgeon until surgery. The method of randomization was concealed envelopes.

ELIGIBILITY:
Inclusion Criteria:

* criteria for bariatric surgery published in 1991 for the National Institutes of Health of the USA.
* age between 18-65 years-old.
* BMI between 40-50 kg/m2
* Obesity for more than 5 years of evolution
* Fail in medical supervised weight loss program
* patient knowing of the mechanism of weight loss after surgery and agreement to collaborate with medical recommendations, diet, medical treatment, as well as the visit established in the follow up program
* patient accepting that surgery objective is not to achieve the ideal weight.
* signed specific informed consent
* women will agree in avoid gestation during one year after surgery

Exclusion Criteria:

* Patients unable to sign the informed consent form because of a mental disorder.
* endocrine diseases causing obesity
* unstable mental disorder, evaluated for a psychiatry MD.
* high anesthetic risk making surgery too risky.
* Malignant neoplasm
* Gastroesophageal reflux disease (GERD) with endoscopic esophagitis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-06; Primary Completion 2019-11 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Hospital Cost in euros | up to 3 months
  Total hospital expenses during admission for the surgery
Length of operation in minutes | 1 day
  Duration of the surgical procedure

SECONDARY OUTCOMES:
weight loss in kilograms | 3 months
  weight of the patient at clinics, 3 months after surgery
weight loss in kilograms | 6 months
  weight of the patient at clinics, 6 months after surgery
weight loss in kilograms | 9 months
  weight of the patient at clinics, 9 months after surgery
weight loss in kilograms | 12 months
  weight of the patient at clinics, 12 months after surgery
weight loss in kilograms | 18 months
  weight of the patient at clinics, 18 months after surgery
weight loss in kilograms | 24 months
  weight of the patient at clinics, 24 months after surgery
weight loss in kilograms | 3 years
  weight of the patient at clinics, 3 years after surgery
weight loss in kilograms | 4 years
  weight of the patient at clinics, 4 years after surgery
weight loss in kilograms | 5 years
  weight of the patient at clinics, 5 years after surgery

OTHER OUTCOMES:
Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment | through study completion an average of 5 year
  Record of any adverse event and/or abnormal laboratory values in relation with the operation performed since the day of the operation to the study completion.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel J Garcia-Oria, MD PhD FACS, Study Chair — Unidad Cirugia Obesidad y Metabolica Hospital Puerta de Hierro
Locations (1):
- Servicio de Cirugía General. Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
The plan is to publish the results of our study in a scientific journal when it be completed, not to publish the individual patient data, just the global data comparing both groups of study.

REFERENCES:
- [Background] Lee WJ, Ser KH, Lee YC, Tsou JJ, Chen SC, Chen JC. Laparoscopic Roux-en-Y vs. mini-gastric bypass for the treatment of morbid obesity: a 10-year experience. Obes Surg. 2012 Dec;22(12):1827-34. doi: 10.1007/s11695-012-0726-9. PMID 23011462
- [Background] Rutledge R. The mini-gastric bypass: experience with the first 1,274 cases. Obes Surg. 2001 Jun;11(3):276-80. doi: 10.1381/096089201321336584. PMID 11433900
- [Background] Lee WJ, Yu PJ, Wang W, Chen TC, Wei PL, Huang MT. Laparoscopic Roux-en-Y versus mini-gastric bypass for the treatment of morbid obesity: a prospective randomized controlled clinical trial. Ann Surg. 2005 Jul;242(1):20-8. doi: 10.1097/01.sla.0000167762.46568.98. PMID 15973097
- [Background] Lee WJ, Lin YH. Single-anastomosis gastric bypass (SAGB): appraisal of clinical evidence. Obes Surg. 2014 Oct;24(10):1749-56. doi: 10.1007/s11695-014-1369-9. PMID 25056233
- [Background] Piche ME, Auclair A, Harvey J, Marceau S, Poirier P. How to choose and use bariatric surgery in 2015. Can J Cardiol. 2015 Feb;31(2):153-66. doi: 10.1016/j.cjca.2014.12.014. Epub 2014 Dec 15. PMID 25661550
- [Background] Ramos AC, Silva AC, Ramos MG, Canseco EG, Galvao-Neto Mdos P, Menezes Mde A, Galvao TD, Bastos EL. Simplified gastric bypass: 13 years of experience and 12,000 patients operated. Arq Bras Cir Dig. 2014;27 Suppl 1(Suppl 1):2-8. doi: 10.1590/s0102-6720201400s100002. PMID 25409956